CLINICAL TRIAL: NCT01466946
Title: Understanding Symptom Recognition and Treatment Decision-making in Hispanic/Latino Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The Sophie Davis School of Biomedical Education The City College of New York (Unknown); City University of New York (Other)
Responsible Party: Sponsor
Other Study IDs: 11-109
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; Hispanic/Latino patients; interviews; 11-109
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- semi-structured interviews: A qualitative study of MSKCC lung cancer patients of Hispanic/Latino descent by collecting retrospective patient narratives to understand the processes that led them to seek medical help when they did, their experiences in seeking and receiving medical guidance, as well as their decisions regarding lung cancer treatment. In addition, we will explore how these patients' representations of lung cancer with its associated risk factors and symptoms affected their treatment decisions.
  Interventions: Behavioral: semi-structured interviews

INTERVENTIONS:
Behavioral: semi-structured interviews — Use semi-structured interview methods to gather narrative data from research participants, as more open-ended interviews allow participants to share information that is most relevant to their own experiences (Patton, 2002; Rubin & Rubin, 2005; Kvale, 1996). Semi-structured interviewing can generate a rich understanding of a participant's life routines, experiences, and attitudes related to a topic of inquiry, and can yield a nuanced and thorough description of a research participant's life story and belief systems.

SUMMARY:
The purpose of the study is to understand why Hispanic/Latino patients with lung cancer are diagnosed later than other groups.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Hispanic/Latino patients with biopsy-proven primary lung cancer treated at MSKCC, including stages of disease I-IV
* 18 years of age or older
* Fluent in English or Spanish
* Patients must reside in the U.S

Exclusion Criteria:

* Spanish-surnamed patients who do not self identify as Hispanic/Latino (e.g., Philippines-born individuals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Self-identified Hispanic/Latino patients with biopsy-proven primary lung cancer treated at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
psychosocial issues | 2 years
  related to lung cancer symptom recognition, delays in lung cancer diagnosis of Hispanic/Latino patients and treatment decision-making processes.
cultural issues | 2 years
  related to lung cancer symptom recognition, delays in lung cancer diagnosis of Hispanic/Latino patients and treatment decision-making processes.

SECONDARY OUTCOMES:
identify obstacles | 2 years
  that have been overcome by Hispanic/Latino lung cancer patients who have succeeded in obtaining access to care at an NCI-designated cancer center, and probe for barriers that these individuals believe still need to be addressed or that they were not successful in surpassing.

CONTACTS AND LOCATIONS:
Overall Officials: William Alago, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm